CLINICAL TRIAL: NCT00814528
Title: Photodynamic Therapy Mediated by Topical Application of 5- ALA for the Treatment of Actinic Keratoses
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study never started due to the Principal Investigator leaving the institution
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15725A
Record Dates: First submitted 2008-12-23; First posted 2008-12-25 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Actinic Keratosis
Keywords: actinic keratosis; skin lesions; 5-ALA; AK; Blu-Light
MeSH Terms: conditions — Keratosis, Actinic | interventions — Fluorouracil; Imiquimod; Therapeutics; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Application of 5-ALA PDT to some lesions on skin with "Blue U" light source (417 nm).
  Interventions: Drug: 5-ALA plus Blu-Light
- 2 (Experimental): 5-FU, Imiquimod or treatment with cryotherapy to lesions on the skin.
  Interventions: Drug: 5-FU, Imiquimod or treatment with cryotherapy

INTERVENTIONS:
Drug: 5-ALA plus Blu-Light — 20% 5-ALA ampoules will be crushed and prepared for application after shaking for 3 minutes. Topical ALA will be applied liberally on skin with extra pressure on lesions. Incubation of ALA will take place for 0-3 hours. Exposure to Blue U light source (417 nm) (DUSA), will be performed for Actinic Keratosis for 15 minutes. Application of combination light sources will be performed when lesions are traced with one pass of Pulsed dye laser (595 nm) (Candela) followed by exposure to Blue U light source for 5-8 minutes pending response.
  Arms: 1
Drug: 5-FU, Imiquimod or treatment with cryotherapy — Cryotherapy will be performed on lesions only every 2 week intervals. Application of Imiquimod will be done on the treated skin area 5 days weekly for 4-6 weeks. 5-FU will be once daily on the treated areas 4- 6 weeks. Responses will be monitored every 2 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to compare the treatment of skin growths called actinic keratoses (AK) with 5-ALA PDT, an FDA-approved treatment, versus treatment with other conventionally used FDA-approved agents such as cryotherapy, Imiquimod, or 5-fluorouracil (5-FU).

ELIGIBILITY:
Inclusion Criteria:

* 18-95 years old
* Diagnosied with actinic keratoses.

Exclusion Criteria:

* Patients who have had Isotretinoin therapy less that 1 year prior to screening.
* Patients who have an adverse reaction to light exposure (for example photo- exacerbated seizures).
* History of porphyria

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Actinic keratosis /incomplete therapy and reoccurence | 18 months

SECONDARY OUTCOMES:
Erythema | 2 weeks post therapy
  Early skin responses 2 weeks post therapy (erythema, scaling, post inflammatory skin changes, fine wrinkling of skin, mottled pigmentation)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Tsoukas, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States